CLINICAL TRIAL: NCT02874521
Title: Effects of Intra-dialytic Low-frequency Electrical Muscle Stimulation and Cycle Training on Cardiorespiratory Function and Muscular Strength: a Pilot Randomized Controlled Trial
Brief Title: Low-frequency Electrical Muscle Stimulation vs Cycle Training During Haemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: Warwick Medical School (Other); Cardiff Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GM118313
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intra-dialytic LF-EMS (Experimental): Performed twice weekly whilst seated on a standard dialysis chair. Delivered by adhesive electrodes in a neoprene garment, applied bilaterally to the quadriceps and hamstrings. Cardiovascular stimulus via rapid, rhythmical, sub-tetanic contractions. Short bursts of four pulses repeatedly delivered by stimulator at a frequency of 4Hz. Current amplitude adjustable from 40 - 200 mA with inbuilt controller. Conducted for one hour at the maximum tolerable intensity. Five minute warm-up and cool down at a lower frequency (3 Hz).
  Interventions: Other: Intra-dialytic LF-EMS
- Intra-dialytic cycle training (Experimental): Semi-recumbent cycling performed twice weekly whilst seated on a standard dialysis chair. Performed for up to one hour per session, initially at a workload (Watts) equivalent to that achieved at 40-60% VO2 reserve during cardiopulmonary exercise test. Exercise intensity regulated using a combination of heart rate and rating of perceived exertion (12-14). Workload adjusted weekly and controlled with a combination of pedal resistance and cadence to provide a personalised exercise prescription. Five minute warm-up and cool down each session.
  Interventions: Other: Intra-dialytic cycle training
- Usual care (No Intervention): Continuation of dialysis treatment without the addition of an intra-dialytic exercise intervention.

INTERVENTIONS:
Other: Intra-dialytic LF-EMS — Electrical muscle stimulation during haemodialysis
  Other Names: Electrical muscle stimulation
  Arms: Intra-dialytic LF-EMS
Other: Intra-dialytic cycle training — Cycle training during haemodialysis
  Arms: Intra-dialytic cycle training

SUMMARY:
The purpose of the trial is to compare the effects of intra-dialytic low-frequency electrical muscle stimulation and intra-dialytic cycling, with usual care haemodialysis without exercise training.

DETAILED DESCRIPTION:
End stage renal disease is associated with reduced functional capacity. Dynamic exercise training i.e. cycling, performed between dialysis sessions or during dialysis (intra-dialytic) can be effective in improving functional capacity and quality of life. However, many patients are unable to engage in intra-dialytic cycling due to limiting comorbidities. Other exercise modalities should be considered. Low-frequency electrical muscle stimulation of the quadriceps is well tolerated and may improve functional capacity in clinical populations.

The trial is a longitudinal, randomised controlled trial. Participants will be randomly allocated to 10 weeks of 1) intra-dialytic low-frequency electrical muscle stimulation, 2) intra-dialytic cycling, or 3) usual care haemodialysis without exercise training. Outcomes will be assessed at baseline and 10 weeks by assessors blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

1. On haemodialysis for at least 3months
2. On 3 times 4 hours of dialysis per week
3. Urea reduction rate of at least 65% during the three months before enrolment
4. Age 18 years or older
5. Able to complete the exercise test and exercise training
6. Able to provide informed consent
7. Life expectancy of more than 6 months according to clinical assessment

Exclusion Criteria:

1. Clinically significant valvular insufficiency
2. Clinically significant dysrythmia
3. Uncontrolled blood pressure: systolic > 160, diastolic >95 during the months before enrolment
4. Excessive fluid accumulation between dialysis sessions (>3 liters), more than twice pulmonary edema over 3 months before enrolment deemed to be due to excess fluid intake
5. Haemoglobin unstable and below 9.0
6. Ischemic cardiac event or intervention in the last 3 months
7. Clinically significant, still active inflammatory or malignant process
8. Pacemaker or cardiac device (contraindicated for bioelectrical impedance)
9. Planned kidney transplant during study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake (VO2peak) | Baseline, 10 weeks
  Cardiopulmonary exercise test

SECONDARY OUTCOMES:
Muscular strength | Baseline, 10 weeks
  Hand held dynamometer - quadriceps strength
Arterial remodelling | Baseline, 10 weeks
  Tonometry - pulse wave velocity
Cardiac remodelling | Baseline, 10 weeks
  Echocardiography - left ventricular volumes
Health related quality of life | Baseline, 10 weeks
  Questionnaire - KDQOL-36

CONTACTS AND LOCATIONS:
Overall Officials: Godon S McGregor, PhD, Study Chair — UHCW NHS Trust
Locations (1):
- University Hospital, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 2021 exceptional surveillance of chronic kidney disease (NICE guideline NG203) [Internet]. London: National Institute for Health and Care Excellence (NICE); 2021 Aug 25. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK576880/ PMID 35077091
- [Background] Heiwe S, Jacobson SH. Exercise training for adults with chronic kidney disease. Cochrane Database Syst Rev. 2011 Oct 5;2011(10):CD003236. doi: 10.1002/14651858.CD003236.pub2. PMID 21975737
- [Background] Bowen TS, Schuler G, Adams V. Skeletal muscle wasting in cachexia and sarcopenia: molecular pathophysiology and impact of exercise training. J Cachexia Sarcopenia Muscle. 2015 Sep;6(3):197-207. doi: 10.1002/jcsm.12043. Epub 2015 Jun 3. PMID 26401465
- [Background] Koufaki P, Mercer TH, Naish PF. Effects of exercise training on aerobic and functional capacity of end-stage renal disease patients. Clin Physiol Funct Imaging. 2002 Mar;22(2):115-24. doi: 10.1046/j.1365-2281.2002.00405.x. PMID 12005153
- [Background] Cheema B, Abas H, Smith B, O'Sullivan A, Chan M, Patwardhan A, Kelly J, Gillin A, Pang G, Lloyd B, Fiatarone Singh M. Randomized controlled trial of intradialytic resistance training to target muscle wasting in ESRD: the Progressive Exercise for Anabolism in Kidney Disease (PEAK) study. Am J Kidney Dis. 2007 Oct;50(4):574-84. doi: 10.1053/j.ajkd.2007.07.005. PMID 17900457
- [Background] Smart NA, Dieberg G, Giallauria F. Functional electrical stimulation for chronic heart failure: a meta-analysis. Int J Cardiol. 2013 Jul 15;167(1):80-6. doi: 10.1016/j.ijcard.2011.12.019. Epub 2012 Jan 10. PMID 22236510
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639